CLINICAL TRIAL: NCT04781517
Title: Development of a Patient-reported Outcome Instrument for Patients With Lumbar Degenerative Disease After Lumbar Fusion
Acronym: DPROIPLDDALF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LDDAFQ-PRO
Record Dates: First submitted 2021-02-18; First posted 2021-03-04 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2021-02

CONDITIONS: Lumbar Spine Degeneration
Keywords: lumbar spine; questionnaire; patient reported outcome measures; quality of life; lumbar fusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Short-segment group: Lumbar degenerative diseases' patients,whose lumbar fixed segments less than 3 was divided into Short-segment group(200).
- Long-segment group: Lumbar degenerative diseases' patients,whose lumbar fixed segments no less than 3 was divided into Long-segment group(200).

SUMMARY:
The commonly used scales (ODI+JOA-29+VAS) lack the assessment of lumbar stiffness, and there is no scale for evaluating lumbar stiffness in China.Based on the Delphi method and the analytic hierarchy process, this study will improve and optimize the quality of life evaluation system for patients with severe degenerative lumbar disease, so as to obtain a concise, practical, and effective patient-reported outcome instrument.

DETAILED DESCRIPTION:
Although lumbar fusion can improve function by correcting deformity,restoring spinal stability,and reducing pain, it also by intention leads to spinal stiffness which can impair function of daily activities.The commonly used scales (ODI+JOA-29+VAS) lack the assessment of lumbar stiffness.Lumbar Stiffness Disability Index (LSDI) has not been used widely, and there is no scale for evaluating lumbar stiffness in China.In addition, even if LSDI is modified, there is still an evaluation dilemma: after lumbar long-segment fixation, the pain and neurological function-related scale scores show that the quality of life is improved, while the lumbar stiffness-related scale scores show that the quality of life is reduced . So overall, is the patient's quality of life improved or decreased? Simply combining these two types of scales cannot explain clearly.

This study can be roughly divided into the following 5 main steps:

Step 1:Collect and sort out the dimensions and exhaustive items that affect the patients' quality of life by systematically reviewing the related literature and a qualitative interview study.

Step 2: Through a cross-sectional survey and experts' meetings, the items is initially optimized, and 35-45 items will be retained.

Step 3: Screen 20-25 excellent items by 2-3 rounds of Delphi method, then use the analytic hierarchy process to determine the weight of each item, so as to establish a initial PRO instrument.

Step 4: Verify the reliability and validity of the initial PRO instrument, and further optimize the initial PRO instrument in order to be used in clinical practice and research.

Step 5: Verify the responsiveness of the initial PRO instrument, calculate the ES, SRM, AUC and MICD values of the initial PRO instrument.

Finally, a novel, concise, practical, and effective PRO instrument for use in degenerative lumbar disease patients will be established.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Lumbar Spine Degeneration
* Plan for or have undergone lumbar fusion
* Be willing to participate in this research

Exclusion Criteria:

* Combined with neurological disease such as Motor neuron disease, Progressive muscular dystrophy, Peripheral neuropathy, Spinal cord disease, et al.
* Combined with severe cervical/thoracic spine disease or other diseases that seriously affect the quality of life
* Suffer lumbar spine trauma after lumbar fusion
* Preoperative cases exclude patients who plan for revision surgery
* Be unwilling to participate in this research

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with lumbar degenerative diseases,planning or undergone their first lumbar fusion,are willing to participate in this research.They have no neurological diseases, severe cervical/thoracic spine disease or other diseases which seriously affect their quality of life, and haven't suffered lumbar trauma after lumbar fusion.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
The Oswestry Disability Index (ODI) | In 7 days before lumbar fusion
  Use the Oswestry Disability Index (ODI) to assess the quality of life of Patients with lumbar degenerative diseases before lumbar fusion.The minimum value of ODI score is 0 and the maximum value is 50. Higher ODI scores mean a worse outcome.
The Japanese Orthopedic Association score(JOA-29) | In 7 days before lumbar fusion
  Use the Japanese Orthopedic Association score(JOA-29) to assess the quality of life of Patients with lumbar degenerative diseases before lumbar fusion.The minimum value of JOA-29 score is 0 and the maximum value is 29. Higher JOA-29 scores mean a better outcome.
The novel PRO instrument | In 7 days before lumbar fusion
  Use the novel PRO instrument to assess the quality of life of Patients with lumbar degenerative diseases before lumbar fusion.The minimum value of the novel PRO instrument score is 0 and the maximum value is 100. Higher the novel PRO instrument scores mean a worse outcome.
The Oswestry Disability Index (ODI) | 6 months after lumbar fusion
  Use the Oswestry Disability Index (ODI) to assess the quality of life of Patients with lumbar degenerative diseases before lumbar fusion.The minimum value of ODI score is 0 and the maximum value is 50. Higher ODI scores mean a worse outcome.
The Japanese Orthopedic Association score(JOA-29) | 6 months after lumbar fusion
  Use the Japanese Orthopedic Association score(JOA-29) to assess the quality of life of Patients with lumbar degenerative diseases before lumbar fusion.The minimum value of JOA-29 score is 0 and the maximum value is 29. Higher JOA-29 scores mean a better outcome.
The novel PRO instrument | 6 months after lumbar fusion
  Use the novel PRO instrument to assess the quality of life of Patients with lumbar degenerative diseases before lumbar fusion.The minimum value of the novel PRO instrument score is 0 and the maximum value is 100. Higher the novel PRO instrument scores mean a worse outcome.
The Oswestry Disability Index (ODI) | 12 months after lumbar fusion
  Use the Oswestry Disability Index (ODI) to assess the quality of life of Patients with lumbar degenerative diseases before lumbar fusion.The minimum value of ODI score is 0 and the maximum value is 50. Higher ODI scores mean a worse outcome.
The Japanese Orthopedic Association score(JOA-29) | 12 months after lumbar fusion
  Use the Japanese Orthopedic Association score(JOA-29) to assess the quality of life of Patients with lumbar degenerative diseases before lumbar fusion.The minimum value of JOA-29 score is 0 and the maximum value is 29. Higher JOA-29 scores mean a better outcome.
The novel PRO instrument | 12 months after lumbar fusion
  Use the novel PRO instrument to assess the quality of life of Patients with lumbar degenerative diseases before lumbar fusion.The minimum value of the novel PRO instrument score is 0 and the maximum value is 100. Higher the novel PRO instrument scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Weishi Li, PhD, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
In order to protect the personal information of patients, there is no plan to make individual participant data (IPD) available to other researchers.